CLINICAL TRIAL: NCT03305588
Title: RAD 1601: Pilot Trial of Frameless Virtual Cone Stereotactic Radiosurgical Thalamotomy for Intractable Tremor and Advanced Functional Connectivity Parcellation of the Thalamus
Brief Title: RAD 1601: EDGE Radiosurgery for Intractable Essential Tremor and Tremor-Dominant Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, John Fiveash, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-160811009
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Essential Tremor; Parkinson Disease
Keywords: essential tremor (ET); stereotactic radiosurgery (SRS); radiosurgery (RS); deep brain stimulation (DBS); Parkinson's Disease (PD); tremor-dominant Parkinson's disease (TDPD)
MeSH Terms: conditions — Essential Tremor; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 130 Gy Radiation & Unframed Virtual Cone (Experimental): 130 Gy Virtual Cone Radiosurgery Unframed (Face Mask)
  Interventions: Device: Unframed Virtual Cone

INTERVENTIONS:
Device: Unframed Virtual Cone — The patient will undergo stereotactic radiosurgery. Radiosurgery is a single non-surgical radiation treatment and will be done as an outpatient procedure. High-energy radiation will be delivered to a small, precise area of the patient's brain using a linear accelerator. A face mask (unframed) will be placed over the patient's face to keep their head from moving during the procedure. During the procedure, the study doctor will confirm the exact location that needs to be treated using x-rays and optical imaging cameras. The face mask will hold the patient's head to prevent it from moving and to focus the x-rays and aim them on a small area in the thalamus of the patient's brain. For most patients, the actual time on the radiosurgery treatment machine is 30 to 60 minutes. The face mask will be removed after the treatment.

SUMMARY:
To determine the efficacy of frameless Virtual Cone Radiosurgical Thalamotomy for medically refractory tremor resulting from either Essential Tremor or Tremor-Dominant Parkinson's Disease with the Fahn-Tolosa-Marin Tremor Rating Scale (FTMTRS) in patients who are not candidates for deep brain stimulation (DBS).

DETAILED DESCRIPTION:
Per the National Institute of Neurological Disorders and Stroke, tremor is an involuntary, rhythmic muscle contraction leading to shaking movements in one or more parts of the body. It is a common movement disorder that most often affects the upper extremities but can also occur in the head, vocal cords, torso, and lower extremities. Tremor may be intermittent or constant. It can be present at rest, during action, or mixed between rest and action.

Tremor can occur at any age but it is most common among middle-aged and older adults; once it occurs, it often progresses over time. This disorder shows no gender predilection. Although tremor is not life threatening, it can be severely disabling, making it difficult or even impossible to perform work and daily life tasks.

Deep parts of the brain that control movements appear to be involved in tremor development. However, most types of tremor have no actual known cause. There are some forms that appear to be inherited and run in families. There are more than 20 types of tremor. Tremor can occur on its own (such as essential tremor (ET) or be associated with other neurological disorders, such as Parkinson's disease (PD).

Tremor is a common symptom of Parkinson's disease. The classification of patients with Parkinson's disease into tremor-dominant and non-tremor subtypes is well established. The pathophysiology of tremor in patients with tremor-dominant Parkinson's disease (TDPD) may be distinct from other their other symptoms, such as bradykinesia, rigidity, and gait and balance symptoms. Importantly, tremor in PD responds less well or can even be highly resistant to dopaminergic treatment than bradykinesia and rigidity. Therefore other treatment strategies may need to be considered.

Essential Tremor (ET) is a common neurologic condition characterized by a tremor that can occur either with posture or action. In the US, there are reported to be as many as 10 million people with essential tremor. A significant subset of patients experience persistent disability and disruption on activities of daily living from tremor and require intervention.

Treatment approach depends on the penetrance of disability into a patient's life, but typically begins with pharmacologic intervention. Patients with disabling tremor refractory to primary and secondary pharmacologic interventions are evaluated for surgical treatment with deep brain stimulation (DBS) or thalamotomy. However, a sizeable subset of these patients are unfavorable candidates for surgery due to medical or neurological co-morbidities. Additionally, a significant subset of patients simply does not wish to undergo the awake craniotomy required for DBS lead placement for tremor. Stereotactic radiosurgery (SRS) thalamotomy is an alternative for those patients. SRS thalamotomy targets the ventral intermediate (VIM) nucleus of the thalamus based on predetermined stereotactic coordinates.

Almost all prior SRS thalamotomy studies performed have used the Leksell Gamma Knife treatment unit and demonstrate that about 80% of properly selected patients respond. The efficacy of Gamma Knife radiosurgery for tremor has been studied prospectively and has been modeled based upon prognostic factors in larger retrospective studies. These studies provide benchmarks for measuring the safety and efficacy of frameless Virtual Cone radiosurgery in this trial. In order for possible frameless Virtual Cone radiosurgery to be a standard of care in the treatment of tremor, additional clinical data is required. This pilot trial of Virtual Cone radiosurgery will assess the safety and efficacy of this treatment. A target of forty patients will be treated to confirm the feasibility of the protocol procedures, efficacy, and safety of the treatment. Secondary endpoints will include quality of life and patient satisfaction. The investigators hypothesize that the recent improvements in LINAC delivery, image guidance, and patient position monitoring will allow a safe frameless procedure that has a high patient satisfaction and low toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with medical refractory essential tremor or tremor-dominant Parkinson's disease that are not candidates for deep brain stimulation (DBS), either by medical/surgical co-morbidities or by choice.
* Patients must have an ECOG status of 0, 1, or 2.
* Patients must be at least 18 years of age.
* All patients must be given written informed consent.

Exclusion Criteria:

* Patients who have had prior radiosurgery or therapeutic brain radiation therapy.
* Patients with medical contra-indications to MRI imaging (e.g. pacemaker).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall tremor reduction proportion evaluated by the Fahn-Tolosa-Marin Tremor Rating Scale (FTMTRS) | From Baseline up to 36 months following completion of radiosurgery
  The Fahn-Tolosa-Marin Tremor Rating Scale evaluation will assess the severity of the patient's tremor and measure the impact on their activities of daily living.

SECONDARY OUTCOMES:
Number of Participants with treatment-related adverse events | From Baseline up to 36 months following completion of radiosurgery
  Based on the assessments of the patient and the responses provided by the patient in questionnaires, the investigators will assess acute and late neurologic toxicities. All adverse events/toxicities will be assessed with the utilization of CTCAE v.4.0.
Changes in resting-state functional MRI (fMRI) and diffusion tensor patterns associated with Radiosurgical thalamotomy | From Baseline up to 36 months following completion of radiosurgery
  Changes will be assessed by resting-state functional MRI (fMRI) to see the impact of radiosurgery ablation on brain function or alteration of function of the ventral intermediate nucleus of the thalamus.
Mean of Quality of Life Scores measured by SF-36 questionnaire | From Baseline up to 36 months following completion of radiosurgery
  Quality of Life (QOL) will be measured by SF-36 questionnaire. This questionnaire consists of 36 questions (items) measuring physical and mental health in relation to 8 health concepts: physical functioning, bodily pain, role of limitations due to physical health problems, role of limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perception. All items are scored so that a high score defines a more favorable health state. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are set at 0 and 100, respectively.
Mean of Quality of Life Scores measured by PROMIS Upper Extremity Questionnaire | From Baseline up to 36 months following completion of radiosurgery
  PROMIS Upper Extremity questionnaire will assess effect of tremor on one's physical function of upper extremity, as well as, effects on activities of daily living.
Patient Satisfaction Scores | 3 Month Follow-Up Visit
  3 months following the completion of radiosurgery, the patient will be asked the following two questions: 1) Would the participant have the radiosurgery procedure again? 2) Would the participant recommend it to friends and family?
Define Targeting Methods within Thalamus based on Structural and Functional Connectivity | From Baseline up to 36 months following completion of radiosurgery
  Compare how well the standard MRI conventional thalamotomy targeting technique (based on predetermined atlas coordinates) matches with advanced MRI-based (functional and structural) mapping of the thalamotomy target.
Mean of Quality of Life Scores measured by the Essential Tremor Rating Assessment Scale (TETRAS) | From Baseline up to 36 months following completion of radiosurgery
  TETRAS scale will assess 9 performance items of examination to create a clinical rating scale for essential tremor. Score is 0-4. Zero being no tremor.

CONTACTS AND LOCATIONS:
Overall Officials: John Fiveash, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham (UAB) Hazelrig-Salter Radiation Oncology Center, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Middlebrooks EH, Popple RA, Greco E, Okromelidze L, Walker HC, Lakhani DA, Anderson AR, Thomas EM, Deshpande HD, McCullough BA, Stover NP, Sung VW, Nicholas AP, Standaert DG, Yacoubian T, Dean MN, Roper JA, Grewal SS, Holland MT, Bentley JN, Guthrie BL, Bredel M. Connectomic Basis for Tremor Control in Stereotactic Radiosurgical Thalamotomy. AJNR Am J Neuroradiol. 2023 Feb;44(2):157-164. doi: 10.3174/ajnr.A7778. Epub 2023 Jan 26. PMID 36702499